CLINICAL TRIAL: NCT00067444
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Fixed Dose Study Evaluating the Efficacy and Safety of Paroxetine CR in Elderly Outpatients Diagnosed With Major Depressive Disorder
Brief Title: Depression Study In Elderly Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29060/874
Record Dates: First submitted 2003-08-19; First posted 2003-08-21 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Depressive Disorder, Major; Major Depressive Disorder (MDD)
Keywords: Elderly; Major Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paroxetine CR

SUMMARY:
Major Depressive Disorder (MDD) Study in Elderly Outpatients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD).
* Current major depressive episode at screen at least 2 months duration.
* Must be at least 60 years of age.

Exclusion Criteria:

* Patients with a primary diagnosis other than MDD.
* Patients with a history of schizophrenia, schizoaffective disorder, bipolar disorder or dementia.
* Patients with a history of brief depressive episodes lasting less than 8 weeks.
* Patients receiving formal psychotherapy within 12 weeks of study.
* Patients who are suicidal.
* Patients who have received electroconvulsive therapy or transcranial magnetic stimulation within 6 months prior to screening.
* Patients with a history or seizure disorders.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2003-06; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the week 10 last observation carried forward endpoint in the 17-item HAM-D total score. | 10 Weeks

SECONDARY OUTCOMES:
Mean change from baseline in HAM-D item 1; Mean change from baseline in the CGI severity of illness score at study endpoint; Percentage of patients with HAM-D total score less than or equal to 7. | 10 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (43):
- United States (43):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, El Centro, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Redlands, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Leesburg, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sebring, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Prairie Village, Kansas
  - GSK Investigational Site, Gaithersburg, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Braintree, Massachusetts
  - GSK Investigational Site, Nashua, New Hampshire
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, Mount Kisco, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Conshohocken, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Pitts CD, Schaefer D, Lipschitz A, Iyengar M: Efficacy and Tolerability of Fixed, Low Dose Paroxetine CR in the Treatment of Depression in the Elderly, Poster No. NR701, presented at the American Psychiatric Association Annual Meeting, May 2005. Available at: www.psych.org
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 29060/874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 29060/874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 29060/874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 29060/874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 29060/874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 29060/874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register